CLINICAL TRIAL: NCT05449977
Title: Evaluation of Physical Activity, Physical Fitness, and Quality of Life in Patients With Schizophrenia Utilized From Community Mental Health Center Services
Brief Title: Evaluation of Physical Activity, Physical Fitness, and Quality of Life in Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/514/227/4
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Physical Activity; Physical fitness; Quality of life
MeSH Terms: conditions — Schizophrenia; Motor Activity | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Schizophrenia: 20 patients with schizophrenia will be conducted
  Interventions: Diagnostic Test: Diagnose

INTERVENTIONS:
Diagnostic Test: Diagnose — First, the participants will be asked to fill out a structured questionnaire containing their sociodemographic characteristics. Then, the 2-minute walk test, the International physical activity questionnaire, the SF-36 short form, and the World health organization quality of life questionnaire will be applied respectively.

SUMMARY:
The aim of this study is to evaluate schizophrenic patients who benefit from community mental health center services in terms of physical activity, physical fitness, and quality of life.

DETAILED DESCRIPTION:
Mental health is defined (according to the World Health Organization) as a state of well-being in which a person can realize his/her abilities, coping with the normal stresses of life, and supporting society by working efficiently and productively. In other words, mental health is a dynamic internal balance that enables individuals to use their diversity of skills in harmony with the universal values of the society. For example, it is the flexibility and ability to cope with negative life experiences and social functioning and the harmonious connection between body and mind. To be more concrete, mental health includes different components of life, for example in terms of relationships, good relationships with friends and family, the ability to talk about feelings. Examples of leisure activities include taking up a hobby, exercising regularly, and routinely taking vacations. It is also important to maintain a lifestyle that consists of having a nutritious and regular diet, not smoking and using over-the-counter drugs, and achieving at least some goals in life.

Mental disorders involve a wide variety of problems. Mental disorders are often characterized by a combination of abnormal thoughts, behaviors, emotions, and relationships with other people. Mental disorders include: depression, drug use disorders, mental disabilities, bipolar disorder and schizophrenia.

Schizophrenia is a chronic mental disorder characterized by the appearance of both positive symptoms such as hallucinations and delusions and negative symptoms such as apathy and withdrawal, repetition of cognitive skills and disorganization. The number of schizophrenic patients in the world is approximately 20 million and this number will continue to increase every year. According to a systematic review of general population studies, the lifetime median prevalence of schizophrenia in Turkey was found to be 8.9 per 1000 people. In addition, schizophrenia patients have irregular self-esteem, inability to maintain social relationships, deterioration in cognitive skills, and sedentary behaviors in their daily lives. Sedentary behavior in patients with schizophrenia will increase the risks of cardiovascular and obstructive pulmonary disease, diabetes mellitus (especially type 2), cancer that can contribute greatly to death and disability. Therefore, it was found that patients with schizophrenia have a shorter life expectancy of 10-20 years compared to the general population.

It has been found that people with schizophrenia are less physically active and less physically fit than the general population. Physical activity means any bodily movement produced by skeletal muscles that results in energy expenditure. Exercise is a subset of physical activity, which is planned, structured and repetitive bodily movements performed to increase and maintain one or more aspects of physical fitness. Physical fitness can be defined as a set of independent qualities associated with the ability to perform physical activities. Components such as cardiorespiratory fitness, muscle strength, muscular endurance and flexibility are more related to health, while components such as coordination and whole-body balance are more related to the performance of physical activities.

There is an inverse relationship between sedentary behavior (related to time spent lying or sitting) and physical activity level in patients with schizophrenia. In addition, physical activity has a direct relationship with physical fitness and physical health in patients with schizophrenia. In addition, one study showed that poor physical activity level and poor physical fitness had a negative effect on the ability of schizophrenia participants to perform activities of daily living performance causes a decrease in the quality of life in these patients. According to the World Health Organization, quality of life is defined as individuals' perceptions of their position in life in the context of the value systems and culture in which they live and in relation to their goals, expectations, standards and concerns. Quality of life is a subjective, multidimensional term defined as a standard level for physical, emotional, material and social well-being.

Community Mental Health Centers are State institutions that provide treatment and rehabilitation services to patients with certain mental health diseases outside the hospital and within the scope of State Hospitals. Community Mental Health Centers (CMHC) were opened in 2011 by the Ministry of Health in Turkey. Patients diagnosed with serious chronic mental disorders such as depression, drug use-related disorders, mental disabilities, bipolar disorder and especially schizophrenia are treated. The aim of these centers is to improve functional recovery, physical activity level and quality of life and integrate it into daily life, society and business life. It consists of a very comprehensive team of different professionals, such as physicians, psychologists, social workers, and nurses.

Schizophrenic patients are treated in a community mental health center with a comprehensive treatment program. The content of the comprehensive rehabilitation program in community mental health centers includes: Psychosocial skills training / occupational treatments such as painting, music, and also these are done according to the patient's condition / psycho-education for patients and their families (information about the disease and treatment, methods of coping with symptoms are explained) training is provided on issues such as illness, crisis management of patients and their relatives), social skills training (patients who cannot participate in social life due to their illness are given training to gain the ability to reorganize human relations) and group treatment is provided for suitable patients.

Evaluation of physical activity levels, physical fitness, and quality of life of patients with schizophrenia is essential to confirm the effectiveness of treatments and care activities at CMHCs and to plan new therapeutic and rehabilitative activities. In one study, they found that the level of physical activity - physical fitness has a positive effect on psychiatric services and can improve the physical health outcomes of people with schizophrenia. They also reveal improvement in psychological and social outcomes in these patients. Therefore, physical activity level and physical fitness are critical parameters of the biopsychosocial approach in recovery-oriented mental health services. In conclusion, our study aims to decide on physical activity, physical fitness and quality of life levels among a group of patients with schizophrenia treated at CMHC and to evaluate the relationship between these three important treatment parameters.

The aim of this study is to evaluate schizophrenic patients who benefit from community mental health center services in terms of physical activity, physical fitness and quality of life. Therefore, given the importance of our study, our findings may contribute to the literature and improvement for mental health systems for people with psychotic disorders, especially schizophrenia. As a result of this study, an evaluation can be made in terms of physical activity, physical fitness and quality of life in schizophrenic patients who receive service from a community mental health center. According to this study, it will be possible to contribute to the effectiveness of treatments and care activities in CMHCs for patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with schizophrenia by a physician according to DSM-5 criteria
* Patients treated at CMHC
* Individuals with schizophrenia who are 18 years or older
* Patients without other comorbid psychiatric disorders
* Patients who can communicate and collaborate
* Patients who agreed to participate in this study and gave informed consent

Exclusion Criteria:

* Those who did not give consent to participate in the study
* Patients with a diagnosis other than schizophrenia
* Pregnancy
* Patients with chronic metabolic diseases such as diabetes, heart problems and cancer

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is planned to include 20 healthy individuals diagnosed with schizophrenia and 20 healthy individuals in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
2 minutes walk test | Up to 6 months
  The American Thoracic Society developed the 2-Minute Walk Test and was officially introduced in 2002 with comprehensive guidelines. The 2-Minute Walk Test measures a person's ability to walk in 2 minutes and their functional capacity (13). In this test, the person walks as fast as possible and without assistance, and then the distance the person walks in 2 minutes is measured. The reliability and validity of the 2 Minute Walk Test (in patients with psychological disorders) was proven in 2019 by Davy Vancampfort et al.
International Physical Activity Questionnaire-Short Form | Up to 6 months
  The International Physical Activity Questionnaire was developed by the international consensus group in 1998. It is used to evaluate the physical activity level of the person, taking into account the last 7 days. Considering the level of physical activity in the IPAQ Short Form, the individual was asked for three specific activity types (walking-moderate and vigorous activity) for the last 7 days. It is also a cost effective method. The reliability and validity of the International Short Form of Physical Activity Questionnaire (IPAQ-SF) was proven by Paul H Lee et al. in 2011 (16).

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Akbuğa Koç, Principal Investigator — Yeditepe Üniversity
Locations (1):
- Ebru Akbuğa Koç, Istanbul, Turkey (Türkiye)